CLINICAL TRIAL: NCT04566679
Title: Butyrate in Children With IBS: Double Blind Placebo Controlled Randomized Clinical Trial
Acronym: BUZIR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Ruggiero Francavilla, Professor, University of Bari
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUZIR2020
Record Dates: First submitted 2020-09-18; First posted 2020-09-28 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Irritable Bowel Syndrome (IBS); Children, Only
Keywords: Irritable Bowel Syndrome (IBS); children
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Butyrate (Experimental): oral butyrate (500mg) once or twice per day
  Interventions: Dietary Supplement: Dibuzin
- Placebo (Placebo Comparator): oral placebo once or twice per day
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Dibuzin — 2-week run-in phase (weeks 1-2) followed by 8-week treatment period (weeks 3-10) and 4-week follow-up phase (weeks 11-14)
  Arms: Butyrate
Dietary Supplement: placebo — 2-week run-in phase (weeks 1-2) followed by 8-week treatment period (weeks 3-10) and 4-week follow-up phase (weeks 11-14)
  Arms: Placebo

SUMMARY:
We will perform a randomized, double-blind, placebo-controlled trial to establish whether calcium butyrate relieves symptoms in children with irritable bowel syndrome (IBS). The direct effects of butyrate on inflammation and GI symptoms will be studied in children with IBS. The design used to study the effects of calcium butyrate will be a double blind randomized placebo-controlled parallel design.

DETAILED DESCRIPTION:
Study plan 2-week run-in phase (weeks 1-2) followed by 8-week treatment period (weeks 3-10) and a 4- week follow-up phase (weeks 11-14).

Randomization Enrolled children will be randomly assigned, with the use of a computer-generated randomization list to receive either oral butyrate (500 mg) or oral placebo once (twice) per day. Placebo and butyrate had the same shape, the placebo's taste, dimension, indication, and appearance.

Data Collection A diary will be given to the parents; on a daily basis, patients will monitor and record the frequency/severity of symptoms and school absence on the diary. To assess the severity of pain, a combination of the self-reported visual analog scale (VAS) and the Faces Pain Scale (FPS) will be used. The 0- to 10-mm VAS scale (0, no pain; 10, worst possible pain) include a horizontal color gradient (green to red) plus a rating. Daily, when asked to evaluate pain, the child would point to a level and trace a line. Assessment will be done coupling the VAS with the FPS, which consists of 6 faces that range from a relaxed face to a face that shows intense pain (von Baeyer CL). GSRS Participants will be asked to fill out the GSRS every 2 weeks during running in, treatment, and follow up (Svedlund).

Compliance To ensure compliance, the investigator will contact the families every 4 weeks to monitor the process of the study.

Adherence will be assessed by counting the number of capsules returned; children who will miss taking more than 20% of the medication will be considered noncompliant.

Fecal Analysis Fecal samples for microbiological analysis will be collected before treatment and at week 10 (end of treatment) and week 14 (4 weeks after discontinuation). Urinary NMR Analysis Urinary samples for NMR analysis will be collected before treatment and at week 10 (end of treatment) and week 14 (4 weeks after discontinuation). This method is described by Lussu et al .

Fecal lactoferrin and calprotectin Fecal calprotectin will be measured using a commercial Fecal Calprotectin Immunoassay kit (Genova Diagnostics, Asheville, NC), respectively, following the manufacturers' instructions.

Sample size calculation To demonstrate an efficacy of butyrate, considering a placebo effect of 20% and a difference in response of at least 35%, keeping a power of the study of 80% and a p of 0,05 we need 23 patients for group that, considering a drop out of 10%, will became 25 per group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IBS according to the Rome IV diagnostic criteria

Exclusion Criteria:

* Presence of any chronic diseases
* Treatment with antibiotics/prebiotics/probiotic/postbiotic in the previous two months
* Diagnosis of another functional GI disease
* Growth failure or others alarming signs of organic conditions
* Previous abdominal surgery

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
butyrate on GI symptoms | daily for 14 weeks
  To assess the severity of pain, a combination of the self-reported visual analog scale (VAS) and the Faces Pain Scale (FPS) will be used. The 0- to 10-mm VAS scale (0, no pain; 10, worst possible pain) include a horizontal color gradient (green to red) plus a rating.
butyrate on GI symptoms | every two weeks for 14 weeks
  Gastrointestinal Symptom Rating Scale (GSRS)

SECONDARY OUTCOMES:
butyrate on inflammation | 14 weeks
  fecal calprotectin and lactoferrin

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Clinica Pediatrica, Bari, Apulia
  - Pediatric Department "B Trambusti" Ospedale Giovanni XXIII Via Amendola 270, Bari, Ba

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gibson P, Rosella O. Interleukin 8 secretion by colonic crypt cells in vitro: response to injury suppressed by butyrate and enhanced in inflammatory bowel disease. Gut. 1995 Oct;37(4):536-43. doi: 10.1136/gut.37.4.536. PMID 7489942
- [Result] Ogawa H, Rafiee P, Fisher PJ, Johnson NA, Otterson MF, Binion DG. Butyrate modulates gene and protein expression in human intestinal endothelial cells. Biochem Biophys Res Commun. 2003 Sep 26;309(3):512-9. doi: 10.1016/j.bbrc.2003.08.026. PMID 12963019
- [Result] Pozuelo M, Panda S, Santiago A, Mendez S, Accarino A, Santos J, Guarner F, Azpiroz F, Manichanh C. Reduction of butyrate- and methane-producing microorganisms in patients with Irritable Bowel Syndrome. Sci Rep. 2015 Aug 4;5:12693. doi: 10.1038/srep12693. PMID 26239401
- [Result] Zhu L, Ma Y, Ye S, Shu Z. Acupuncture for Diarrhoea-Predominant Irritable Bowel Syndrome: A Network Meta-Analysis. Evid Based Complement Alternat Med. 2018 May 27;2018:2890465. doi: 10.1155/2018/2890465. eCollection 2018. PMID 29977312
- [Result] Banasiewicz T, Krokowicz L, Stojcev Z, Kaczmarek BF, Kaczmarek E, Maik J, Marciniak R, Krokowicz P, Walkowiak J, Drews M. Microencapsulated sodium butyrate reduces the frequency of abdominal pain in patients with irritable bowel syndrome. Colorectal Dis. 2013 Feb;15(2):204-9. doi: 10.1111/j.1463-1318.2012.03152.x. PMID 22738315
- [Result] von Baeyer CL. Children's self-reports of pain intensity: scale selection, limitations and interpretation. Pain Res Manag. 2006 Autumn;11(3):157-62. doi: 10.1155/2006/197616. PMID 16960632
- [Result] Svedlund J, Sjodin I, Dotevall G. GSRS--a clinical rating scale for gastrointestinal symptoms in patients with irritable bowel syndrome and peptic ulcer disease. Dig Dis Sci. 1988 Feb;33(2):129-34. doi: 10.1007/BF01535722. PMID 3123181
- [Result] Lussu M, Noto A, Masili A, Rinaldi AC, Dessi A, De Angelis M, De Giacomo A, Fanos V, Atzori L, Francavilla R. The urinary 1 H-NMR metabolomics profile of an italian autistic children population and their unaffected siblings. Autism Res. 2017 Jun;10(6):1058-1066. doi: 10.1002/aur.1748. Epub 2017 Mar 11. PMID 28296209
- [Result] De Angelis M, Piccolo M, Vannini L, Siragusa S, De Giacomo A, Serrazzanetti DI, Cristofori F, Guerzoni ME, Gobbetti M, Francavilla R. Fecal microbiota and metabolome of children with autism and pervasive developmental disorder not otherwise specified. PLoS One. 2013 Oct 9;8(10):e76993. doi: 10.1371/journal.pone.0076993. eCollection 2013. PMID 24130822
- [Derived] Cristofori F, Calabrese FM, Iacobellis I, Santamaria M, Celano G, Ferrocino I, Di Sabato E, Pergola R, Dargenio VN, Paulucci L, De Angelis M, Francavilla R. Calcium butyrate efficacy in pediatric irritable bowel syndrome: Randomized placebo-controlled multiomics-based clinical trial. J Pediatr Gastroenterol Nutr. 2025 Sep;81(3):551-561. doi: 10.1002/jpn3.70154. Epub 2025 Jul 9. PMID 40635319